CLINICAL TRIAL: NCT06288737
Title: Exploring Enrollment and Engagement Trends in Individuals Managing Keratoconus: A Comprehensive Examination of Data on Keratoconus Clinical Trials
Brief Title: Assessing Patient Engagement in Keratoconus Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 54335073
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Keratoconus
Keywords: keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the influences behind patient choices regarding involvement, discontinuation, or re-engagement in keratoconus clinical trials. Uncovering these factors is essential to enhance the relevance and efficacy of future research endeavors.

In essence, this trial aims to deepen understanding of the factors influencing participation in keratoconus clinical trials. Elevating participation rates could expedite the development of innovative treatments for this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Aged ≥ 18 years old
* No prior treatment for keratoconus

Exclusion Criteria:

* Participant is actively receiving study therapy in another
* Inability to provide written informed consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with keratoconus who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in a keratoconus clinical trial | 3 months
Number of keratoconus patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moran S, Gomez L, Zuber K, Gatinel D. A Case-Control Study of Keratoconus Risk Factors. Cornea. 2020 Jun;39(6):697-701. doi: 10.1097/ICO.0000000000002283. PMID 32040008
- [Background] Kandel H, Pesudovs K, Nguyen V, Chen JY, Poon A, Mills R, Watson SL. Patient-Reported Outcomes in Keratoconus: A Save Sight Keratoconus Registry Study. Cornea. 2023 May 1;42(5):590-597. doi: 10.1097/ICO.0000000000003119. Epub 2022 Aug 24. PMID 36036705
- [Background] Aiello F, Gallo Afflitto G, Ceccarelli F, Garzione F, Pocobelli G, Pinci C, Di Lorenzo G, Siracusano A, Nucci C. Keratoconus and Personality Traits: A Case-Control Study. Cornea. 2024 Feb 1;43(2):237-244. doi: 10.1097/ICO.0000000000003284. Epub 2023 Apr 5. PMID 37018764

DOCUMENTS (1):
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT06288737/ICF_000.pdf